CLINICAL TRIAL: NCT03823300
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab in Patients With Neovascular Age-Related Macular Degeneration (LUCERNE)
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab in Participants With Neovascular Age-Related Macular Degeneration (LUCERNE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR40844; 2018-004042-42 (EudraCT Number)
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Wet Macular Degeneration
Keywords: AMD; nAMD; neovascular age-related macular degeneration; choroidal neovascularization secondary to age-related macular degeneration
MeSH Terms: conditions — Wet Macular Degeneration | interventions — faricimab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Faricimab (Experimental)
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- Arm B: Aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered by intravitreal injection into the study eye at intervals as specified in the study protocol.
  Other Names: VABYSMO™; RO6867461; RG7716
  Arms: Arm A: Faricimab
Drug: Aflibercept — Aflibercept will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by once every 8 weeks (Q8W).
  Other Names: Eylea
  Arms: Arm B: Aflibercept
Procedure: Sham Procedure — The sham is a procedure that mimics an intravitreal injection, but involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It will be administered to participants in both treatment arms at applicable visits to maintain masking.

SUMMARY:
This study will evaluate the efficacy, safety, durability, and pharmacokinetics of faricimab administered at intervals as specified in the protocol, compared with aflibercept once every 8 weeks (Q8W), in participants with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve choroidal neovascularization (CNV) secondary to age-related macular degeneration (nAMD) in the study eye
* Ability to comply with the study protocol, in the investigator's judgment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive measures that result in failure rate <1% per year during the treatment period and for at least 3 months after the final dose of study treatment
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* Uncontrolled blood pressure, defined as systolic blood pressure >180 millimeters of mercury (mmHg) and/or diastolic blood pressure >100 mmHg while a patient is at rest on Day 1
* Pregnancy or breastfeeding, or intention to become pregnant during the study
* CNV due to causes other than AMD in the study eye
* Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid in the study eye
* Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study
* Uncontrolled glaucoma in the study eye
* Any prior or concomitant treatment for CNV or vitreomacular-interface abnormalities in the study eye
* Prior IVT administration of faricimab in either eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active ocular inflammation or suspected or active ocular or periocular infection in either eye
* Other protocol-specified exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (137):
- United States (41):
  - Associated Retina Consultants, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retinal Consultants Med Group, Sacramento, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Colorado Retina Associates, PC, Golden, Colorado
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Prairie Retina Center, Springfield, Illinois
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Retina Specialists, Towson, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - VitreoRetinal Surgery, PLLC., Minneapolis, Minnesota
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - Island Retina, Shirley, New York
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - The Ohio State University Havener Eye Institute, Columbus, Ohio
  - Midwest Retina, Dublin, Ohio
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Center of Texas, Grapevine, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, PLLC, Murray, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Pacific Northwest Retina, Silverdale, Washington
- Argentina (7):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Fundacion Zambrano, CABA
  - Centro Oftalmológico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Oftar, Mendoza
  - Grupo Laser Vision, Rosario
- Australia (9):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Marsden Eye Research Centre, Parramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Austria (2):
  - LKH-Univ.Klinikum Graz, Graz
  - Medizinische Universität Wien, Vienna
- Brazil (2):
  - Hospital de Olhos de Aparecida - HOA, Aparecida de Goiânia, Goiás
  - Universidade Federal de Sao Paulo - UNIFESP*X, São Paulo, São Paulo
- Bulgaria (2):
  - Specialized Hospital for Active Treatment of Eye Diseases Zora, Sofia
  - Pentagram Eye Hospital (Medical Center "Pentagram"), Sofia
- China (15):
  - Beijing Friendship Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Southwest Hospital , Third Military Medical University, Chongqing
  - Army Medical Center of PLA(Daping Hospital), Chongqing
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - The Affiliated Eye Hospital of Nanjing Medical University, Nanjing
  - Shanghai First People's Hospital, Shanghai
  - He Eye Specialist Shenyang Hospital, Shenyang
  - Tianjin Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Wuxi No.2 People's Hospital, Wuxi
- Denmark (2):
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Sjællands Universitetshospital, Roskilde, Roskilde
- France (9):
  - Chi De Creteil, Créteil
  - Pole Vision Val d'Ouest, Écully
  - Hopital de la croix rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - CHU Nantes - Hôtel Dieu, Nantes
  - Centre Odeon, Paris
  - Hopital Lariboisiere, Paris
  - Centre Ophtalmologique, Paris
  - Centres Ophtalmologique St Exupéry, Saint-Cyr-sur-Loire
- Germany (4):
  - Universitätsklinikum Köln, Cologne
  - Universitätkslinikum Düsseldorf, Augenklinik, Düsseldorf
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster, Münster
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - Hong Kong Eye Hospital, Mong Kok
- Hungary (3):
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Szegedi Tudományegyetem ÁOK, Szeged
- Italy (6):
  - Fondazione Ptv Policlinico Tor Vergata Di Roma, Rome, Lazio
  - UNIVERSITA' DEGLI STUDI DI GENOVA - Di.N.O.G., Genoa, Liguria
  - Asst Fatebenefratelli Sacco, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Nuovo Ospedale S. Chiara - A.O.U.P Presidio Ospedaliero di Cisanello, Pisa, Tuscany
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Veneto
- Poland (4):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzia? Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Caminomed, Tarnowskie Góry
- Portugal (2):
  - Centro Hospitalar E Universitário de Coimbra EPE - Serviço Oftalmologia, Coimbra
  - Hospital de Sao Joao, Porto
- Russia (4):
  - Intersec Research and Technology Complex ?Eye Microsurgery? n.a. S.N. Fyodorov, Cheboksary, Mariy-El Republic
  - 1 Saint-Petersburg St. Med. University named after academician I.P.Pavlov, Saint Petersburg, Sankt-Peterburg
  - ?Intersec. Research and Technology Complex ?Eye Microsurgery? n a Fyodorov Irkutsk branch, Irkutsk
  - ?Intersec Research and Technology Complex Eye Microsurgery n a Fyodorov Novosibirsk Branch, Novosibirsk
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore Eye Research Institute, Singapore
- South Korea (8):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Nune Eye Hospital, Seoul
  - Asan Medical Center., Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Institut de la Macula i la retina, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Turkey (Türkiye) (4):
  - Hacettepe University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Gazi University Faculty of Medicine, Ankara
  - Ege University Medical Faculty, Izmir

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Result] Khanani AM, Kotecha A, Chang A, Chen SJ, Chen Y, Guymer R, Heier JS, Holz FG, Iida T, Ives JA, Lim JI, Lin H, Michels S, Quezada Ruiz C, Schmidt-Erfurth U, Silverman D, Singh R, Swaminathan B, Willis JR, Tadayoni R; TENAYA and LUCERNE Investigators. TENAYA and LUCERNE: Two-Year Results from the Phase 3 Neovascular Age-Related Macular Degeneration Trials of Faricimab with Treat-and-Extend Dosing in Year 2. Ophthalmology. 2024 Aug;131(8):914-926. doi: 10.1016/j.ophtha.2024.02.014. Epub 2024 Feb 19. PMID 38382813
- [Derived] Takahashi K, Cheung CMG, Iida T, Lai TYY, Ohji M, Yanagi Y, Kawano M, Ohsawa S, Suzuki T, Kotecha A, Lin H, Patel V, Swaminathan B, Lee WK; TENAYA, LUCERNE Investigators. Efficacy, durability, and safety of faricimab in patients from Asian countries with neovascular age-related macular degeneration: 1-Year subgroup analysis of the TENAYA and LUCERNE trials. Graefes Arch Clin Exp Ophthalmol. 2023 Nov;261(11):3125-3137. doi: 10.1007/s00417-023-06071-8. Epub 2023 Jun 9. PMID 37294433
- [Derived] Khanani AM, Guymer RH, Basu K, Boston H, Heier JS, Korobelnik JF, Kotecha A, Lin H, Silverman D, Swaminathan B, Willis JR, Yoon YH, Quezada-Ruiz C. TENAYA and LUCERNE: Rationale and Design for the Phase 3 Clinical Trials of Faricimab for Neovascular Age-Related Macular Degeneration. Ophthalmol Sci. 2021 Nov 17;1(4):100076. doi: 10.1016/j.xops.2021.100076. eCollection 2021 Dec. PMID 36246941
- [Derived] Heier JS, Khanani AM, Quezada Ruiz C, Basu K, Ferrone PJ, Brittain C, Figueroa MS, Lin H, Holz FG, Patel V, Lai TYY, Silverman D, Regillo C, Swaminathan B, Viola F, Cheung CMG, Wong TY; TENAYA and LUCERNE Investigators. Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE): two randomised, double-masked, phase 3, non-inferiority trials. Lancet. 2022 Feb 19;399(10326):729-740. doi: 10.1016/S0140-6736(22)00010-1. Epub 2022 Jan 24. PMID 35085502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1012 patients were screened, 354 of whom failed screening, most commonly due to not meeting inclusion criteria. A total of 658 treatment-naive patients with nAMD were randomized 1:1 into the study: 331 to the faricimab arm and 327 to the aflibercept arm.
Groups:
- Arm A: Faricimab: Participants randomized to Arm A received 6 mg of faricimab intravitreally (IVT) once every 4 weeks (Q4W) up to Week 12 (4 injections). At Week 20, protocol-defined assessment of disease activity required Arm A participants with active disease to be treated with a once every 8 weeks (Q8W) dosing regimen of 6 mg of faricimab IVT (i.e., injections at Weeks 20, 28, 36, 44, 52, and 60). A second protocol-defined assessment of disease activity at Week 24 required Arm A participants with active disease (excluding those with active disease at Week 20) to be treated with a once every 12 weeks (Q12W) dosing regimen of 6 mg of faricimab IVT (i.e., injections at Weeks 24, 36, 48, and 60). Participants receiving faricimab who did not have active disease according to the protocol-defined criteria at Week 20 and Week 24 were treated with 6 mg of faricimab IVT once every 16 weeks (Q16W) (i.e., injections at Weeks 28, 44, and 60). From Week 60 (when all Arm A participants were scheduled to receive study drug) to Week 108, Arm A participants were to be treated according to a personalized treatment interval (PTI) dosing regimen (Q8W, Q12W, or Q16W).
- Arm B: Aflibercept: Participants randomized to the active comparator (Arm B) received a 2-mg dose of aflibercept that was administered intravitreally (IVT) Q8W, after 3 consecutive monthly doses during the 108-week treatment period. Participants were to receive 15 IVT injections of aflibercept during the 108-week treatment period comprising three initiating injections (2 mg of aflibercept Q4W to Week 8), followed by 12 maintenance injections (2 mg of aflibercept Q8W at Weeks 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, and 104).
Period: Overall Study
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Started (Intent-to-Treat (ITT) Population) | 331 | 327
Received at Least One Dose of Study Drug (Safety Population) | 331 | 326
Completed up to Week 48 (Primary Completion Date Cutoff) | 321 | 309
Completed | 297 | 273
Not Completed | 34 | 54
Not completed — Withdrawal by Subject | 16 | 22
Not completed — Death | 10 | 14
Not completed — Adverse Event | 3 | 5
Not completed — Physician Decision | 1 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Not Eligible | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept | Total
Number analyzed (Participants) | 331 | 327 | 658
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.8 (8.4) | 76.1 (8.6) | 75.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 188 | 391
  Male | 128 | 139 | 267
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 46 | 81
  Not Hispanic or Latino | 287 | 274 | 561
  Unknown or Not Reported | 9 | 7 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 278 | 270 | 548
  Asian | 38 | 34 | 72
  Unknown | 12 | 17 | 29
  Black or African American | 2 | 5 | 7
  American Indian or Alaska Native | 1 | 0 | 1
  Multiple | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States and Canada | 135 | 132 | 267
  Asia | 35 | 33 | 68
  Rest of the World | 161 | 162 | 323
Number of Participants by the Eye (Right or Left) Chosen as the Study Eye [Count of Participants; unit: Participants]
  Right Eye | 168 | 170 | 338
  Left Eye | 163 | 157 | 320
Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye [Mean (Standard Deviation); unit: ETDRS Letters] — Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
  ETDRS Letters | 58.7 (14.0) | 58.9 (13.3) | 58.8 (13.6)
Number of Participants by the BCVA Letter Score Categories in the Study Eye [Count of Participants; unit: Participants]
  ≥74 Letters | 45 | 39 | 84
  73 to 55 Letters | 181 | 183 | 364
  ≤54 Letters | 105 | 105 | 210
Number of Participants by the Low Luminance Deficit (LLD) Letter Score Categories in the Study Eye [Count of Participants; unit: Participants]
  <33 Letters | 238 | 234 | 472
  ≥33 Letters | 89 | 93 | 182
  Missing/Invalid | 4 | 0 | 4
Choroidal Neovascularization (CNV) Lesion Type in the Study Eye by Fundus Fluorescein Angiography [Count of Participants; unit: Participants]
  Occult | 171 | 140 | 311
  Classic | 98 | 109 | 207
  Minimally Classic | 30 | 31 | 61
  Retinal Angiomatous Proliferation (RAP) | 14 | 15 | 29
  Predominantly Classic | 6 | 16 | 22
  Polypoidal Choroidal Vasculopathy (PCV) | 5 | 8 | 13
  Missing | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The Mixed Model of Repeated Measures (MMRM) analysis adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), baseline BCVA (≥74, 73-55, and ≤54 letters), baseline LLD (<33 and ≥33 letters), and region (U.S. and Canada, Asia, and rest of the world). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded from analysis. 95% CI is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 48
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
ETDRS Letters | 6.6 [5.3 to 7.8] | 6.6 [5.3 to 7.8]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; The null hypothesis, H0: μ(faricimab) - μ(aflibercept) ≤-4 letters; the alternative hypothesis, Ha: μ(faricimab) - μ(aflibercept) >-4 letters. A sample size of approximately 320 participants in each arm provided greater than 90% power to show non-inferiority of faricimab to aflibercept in the change from baseline BCVA averaged over Weeks 40, 44, and 48 in the ITT population, using a non-inferiority margin of 4 letters at the one-sided 0.02485 significance level; Test type: Non-Inferiority — If the lower bound of a two-sided 95.03% confidence interval (CI) for the difference in adjusted means of the two treatments (faricimab minus aflibercept) is greater than -4 letters (the non-inferiority margin), then faricimab is considered non-inferior to aflibercept; Adjusted mean difference = 0.0, 95% CI 2-sided [-1.7 to 1.8], Standard Error of Mean 0.91 — The treatment difference in adjusted means of change from baseline BCVA is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept. MMRM adjustments are listed in the outcome measure description

2. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 1
Time Frame: From Baseline through Week 60
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
ETDRS Letters | 6.6 [5.3 to 7.9] | 7.1 [5.8 to 8.4]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in Adjusted Means at Weeks 52-60; Test type: Other; Adjusted mean difference = -0.6, 95% CI 2-sided [-2.4 to 1.3], Standard Error of Mean 0.93 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Over Time
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, and 112
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
ETDRS Letters
  Week 4 | 5.1 [4.2 to 5.9] | 4.3 [3.5 to 5.2]
  Week 8 | 6.0 [5.1 to 6.9] | 5.8 [4.9 to 6.8]
  Week 12 | 7.0 [6.1 to 8.0] | 6.4 [5.4 to 7.4]
  Week 16 | 6.7 [5.6 to 7.7] | 6.4 [5.4 to 7.4]
  Week 20 | 7.0 [5.9 to 8.1] | 6.8 [5.7 to 7.9]
  Week 24 | 7.0 [5.8 to 8.1] | 6.5 [5.4 to 7.6]
  Week 28 | 7.1 [5.9 to 8.2] | 6.8 [5.6 to 7.9]
  Week 32 | 7.2 [6.0 to 8.3] | 6.9 [5.7 to 8.0]
  Week 36 | 6.7 [5.5 to 7.9] | 6.8 [5.6 to 8.0]
  Week 40 | 6.8 [5.5 to 8.1] | 6.7 [5.4 to 8.0]
  Week 44 | 6.5 [5.3 to 7.8] | 6.4 [5.2 to 7.7]
  Week 48 | 6.5 [5.1 to 7.8] | 6.4 [5.0 to 7.7]
  Week 52 | 6.4 [5.1 to 7.7] | 6.9 [5.5 to 8.3]
  Week 56 | 7.1 [5.7 to 8.4] | 7.4 [6.0 to 8.7]
  Week 60 | 6.3 [4.9 to 7.7] | 6.9 [5.5 to 8.3]
  Week 64 | 6.5 [5.1 to 8.0] | 6.1 [4.7 to 7.6]
  Week 68 | 6.2 [4.8 to 7.6] | 6.7 [5.3 to 8.1]
  Week 72 | 6.4 [4.9 to 7.8] | 6.2 [4.8 to 7.7]
  Week 76 | 6.4 [4.9 to 7.9] | 6.0 [4.6 to 7.5]
  Week 80 | 5.9 [4.4 to 7.4] | 5.6 [4.1 to 7.2]
  Week 84 | 5.9 [4.3 to 7.5] | 5.8 [4.2 to 7.3]
  Week 88 | 5.6 [4.1 to 7.1] | 5.4 [3.9 to 7.0]
  Week 92 | 5.7 [4.2 to 7.2] | 5.4 [3.9 to 7.0]
  Week 96 | 5.4 [3.9 to 7.0] | 5.5 [3.9 to 7.0]
  Week 100 | 5.2 [3.6 to 6.8] | 4.9 [3.3 to 6.5]
  Week 104 | 5.0 [3.4 to 6.6] | 5.3 [3.7 to 6.9]
  Week 108 | 5.2 [3.5 to 6.8] | 5.4 [3.7 to 7.0]
  Week 112 | 4.8 [3.2 to 6.5] | 4.8 [3.1 to 6.5]

4. Secondary Outcome: Percentage of Participants Gaining Greater Than or Equal to (≥)15, ≥10, ≥5, or ≥0 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Participants with at least one non-missing, valid assessment at Weeks 40, 44, or 48 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 302 | 291
Percentage of participants
  Gaining ≥15 Letters | 20.2 [15.9 to 24.6] | 22.2 [17.7 to 26.8]
  Gaining ≥10 Letters | 39.2 [34.1 to 44.4] | 35.8 [30.6 to 40.9]
  Gaining ≥5 Letters | 60.5 [55.2 to 65.7] | 59.4 [53.9 to 64.9]
  Gaining ≥0 Letters | 82.2 [77.9 to 86.4] | 79.1 [74.5 to 83.6]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥15 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -2.0, 95% CI 2-sided [-8.3 to 4.3] — The treatment difference in CMH weighted percentage of participants gaining ≥15 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 2: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥10 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 3.4, 95% CI 2-sided [-3.9 to 10.7] — The treatment difference in CMH weighted percentage of participants gaining ≥10 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 3: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥5 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 1.0, 95% CI 2-sided [-6.6 to 8.6] — The treatment difference in CMH weighted percentage of participants gaining ≥5 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 4: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥0 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 3.1, 95% CI 2-sided [-3.1 to 9.3] — The treatment difference in CMH weighted percentage of participants gaining ≥0 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

5. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 4
Time Frame: Baseline, average of Weeks 52, 56, and 60
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Participants with at least one non-missing, valid assessment at Weeks 52, 56, or 60 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 289 | 276
Percentage of participants | 22.6 [18.1 to 27.1] | 23.7 [19.1 to 28.4]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 52-60; Test type: Other; Difference in CMH Weighted Percentage = -1.2, 95% CI 2-sided [-7.7 to 5.3] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA in the Study Eye Over Time
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: as for outcome 3
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. At a given timepoint, the number analyzed includes participants with a non-missing, valid assessment at that timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 10.5 [7.2 to 13.7] | 9.5 [6.4 to 12.6]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 13.9 [10.3 to 17.5] | 13.5 [10.0 to 17.1]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 17.7 [13.7 to 21.6] | 17.2 [13.3 to 21.1]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 17.3 [13.3 to 21.3] | 17.7 [13.6 to 21.8]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 20.2 [15.9 to 24.4] | 20.2 [15.9 to 24.4]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 19.3 [14.9 to 23.6] | 18.9 [14.6 to 23.3]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 23.7 [19.1 to 28.3] | 20.8 [16.1 to 25.4]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 22.6 [18.0 to 27.2] | 19.5 [15.1 to 23.9]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 22.2 [17.7 to 26.6] | 20.6 [16.1 to 25.0]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 23.7 [19.0 to 28.3] | 25.4 [20.6 to 30.1]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 21.5 [17.1 to 26.0] | 22.4 [17.7 to 27.1]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 22.3 [17.7 to 26.9] | 23.1 [18.3 to 27.8]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 22.7 [18.1 to 27.2] | 23.4 [18.7 to 28.1]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 25.9 [21.1 to 30.7] | 27.0 [22.0 to 32.0]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 22.6 [18.1 to 27.1] | 25.8 [20.9 to 30.7]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 25.4 [20.6 to 30.2] | 21.2 [16.5 to 25.9]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 24.5 [19.7 to 29.3] | 24.9 [20.0 to 29.8]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 22.6 [17.9 to 27.2] | 27.1 [22.0 to 32.1]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 22.1 [17.4 to 26.8] | 24.9 [20.1 to 29.8]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 22.9 [18.1 to 27.7] | 25.8 [20.8 to 30.7]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 23.7 [18.9 to 28.5] | 25.6 [20.6 to 30.6]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 24.1 [19.3 to 29.0] | 24.4 [19.5 to 29.3]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 22.5 [17.8 to 27.2] | 24.8 [19.9 to 29.8]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 25.7 [20.8 to 30.6] | 25.5 [20.5 to 30.6]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 24.8 [19.9 to 29.8] | 23.1 [18.3 to 28.0]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 22.5 [17.7 to 27.3] | 24.6 [19.6 to 29.5]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 21.6 [16.8 to 26.3] | 22.3 [17.5 to 27.1]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 25.2 [20.3 to 30.1] | 22.5 [17.8 to 27.1]

7. Secondary Outcome: Percentage of Participants Gaining ≥10 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 24.2 [19.8 to 28.7] | 22.1 [17.7 to 26.5]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 32.4 [27.5 to 37.2] | 28.7 [24.1 to 33.4]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 34.2 [29.3 to 39.1] | 34.6 [29.5 to 39.7]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 35.3 [30.3 to 40.4] | 34.2 [29.2 to 39.3]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 37.8 [32.7 to 42.9] | 34.3 [29.2 to 39.4]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 39.2 [33.8 to 44.5] | 35.2 [29.9 to 40.5]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 40.5 [35.1 to 45.8] | 36.0 [30.5 to 41.4]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 40.5 [35.1 to 46.0] | 35.0 [29.7 to 40.3]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 38.9 [33.6 to 44.2] | 38.9 [33.5 to 44.3]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 40.9 [35.5 to 46.3] | 39.3 [34.0 to 44.7]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 42.3 [36.8 to 47.8] | 39.5 [34.1 to 45.0]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 41.0 [35.5 to 46.5] | 38.6 [33.2 to 43.9]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 44.2 [38.8 to 49.7] | 42.1 [36.6 to 47.6]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 44.2 [38.8 to 49.7] | 43.6 [38.1 to 49.2]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 43.1 [37.6 to 48.6] | 42.4 [36.8 to 47.9]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 44.0 [38.5 to 49.5] | 41.1 [35.4 to 46.8]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 40.1 [34.7 to 45.5] | 40.7 [35.3 to 46.2]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 42.0 [36.5 to 47.4] | 38.9 [33.4 to 44.3]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 42.2 [36.7 to 47.8] | 40.7 [35.1 to 46.2]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 44.2 [38.6 to 49.9] | 41.9 [36.2 to 47.6]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 42.7 [37.2 to 48.3] | 41.4 [35.6 to 47.2]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 40.3 [34.8 to 45.9] | 39.4 [33.7 to 45.1]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 42.1 [36.5 to 47.8] | 41.0 [35.3 to 46.7]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 41.1 [35.5 to 46.7] | 39.1 [33.3 to 45.0]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 40.2 [34.6 to 45.7] | 34.6 [29.0 to 40.1]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 44.0 [38.3 to 49.7] | 36.2 [30.5 to 41.9]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 41.7 [36.0 to 47.4] | 38.0 [32.2 to 43.8]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 41.3 [35.7 to 47.0] | 35.0 [29.6 to 40.5]

8. Secondary Outcome: Percentage of Participants Gaining ≥5 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 47.8 [42.6 to 53.0] | 47.5 [42.2 to 52.8]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 56.8 [51.6 to 62.0] | 54.6 [49.3 to 59.8]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 63.9 [58.9 to 68.9] | 57.6 [52.3 to 62.9]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 61.7 [56.5 to 66.8] | 59.6 [54.3 to 64.9]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 64.1 [59.0 to 69.2] | 60.9 [55.6 to 66.3]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 62.2 [56.8 to 67.6] | 60.2 [54.7 to 65.7]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 63.6 [58.2 to 68.9] | 60.5 [54.8 to 66.2]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 63.3 [58.0 to 68.7] | 60.1 [54.6 to 65.6]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 61.4 [56.0 to 66.9] | 60.4 [54.9 to 65.9]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 63.5 [58.1 to 68.9] | 60.9 [55.5 to 66.4]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 60.1 [54.6 to 65.6] | 62.3 [56.7 to 67.8]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 60.0 [54.5 to 65.6] | 63.5 [57.9 to 69.1]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 63.5 [58.1 to 69.0] | 67.2 [61.7 to 72.6]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 64.1 [58.7 to 69.5] | 66.5 [61.0 to 72.0]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 61.6 [56.1 to 67.2] | 65.5 [59.9 to 71.0]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 65.2 [59.8 to 70.6] | 63.1 [57.5 to 68.8]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 63.0 [57.4 to 68.5] | 64.0 [58.5 to 69.6]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 64.1 [58.6 to 69.6] | 66.6 [60.9 to 72.2]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 63.9 [58.2 to 69.6] | 58.7 [53.0 to 64.4]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 63.3 [57.7 to 68.9] | 62.3 [56.6 to 67.9]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 61.6 [56.1 to 67.2] | 64.3 [58.6 to 70.1]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 62.6 [57.1 to 68.1] | 60.7 [54.9 to 66.5]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 62.7 [57.1 to 68.3] | 58.3 [52.6 to 64.0]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 61.3 [55.6 to 67.0] | 61.0 [55.1 to 67.0]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 61.7 [56.1 to 67.3] | 56.9 [50.9 to 62.9]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 60.3 [54.6 to 66.0] | 59.3 [53.3 to 65.3]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 62.4 [56.8 to 68.0] | 58.0 [51.8 to 64.1]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 59.9 [54.2 to 65.6] | 59.4 [53.4 to 65.3]

9. Secondary Outcome: Percentage of Participants Gaining ≥0 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 80.5 [76.3 to 84.7] | 74.2 [69.5 to 78.9]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 82.3 [78.3 to 86.3] | 80.3 [76.0 to 84.5]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 84.1 [80.3 to 88.0] | 81.0 [76.8 to 85.1]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 82.6 [78.5 to 86.6] | 83.0 [78.9 to 87.0]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 84.8 [80.9 to 88.6] | 83.1 [79.1 to 87.2]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 82.8 [78.6 to 86.9] | 82.0 [77.6 to 86.4]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 82.7 [78.5 to 86.8] | 83.0 [78.7 to 87.4]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 80.3 [75.9 to 84.7] | 82.2 [77.8 to 86.5]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 81.2 [76.8 to 85.6] | 76.5 [71.7 to 81.3]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 82.0 [77.6 to 86.3] | 77.6 [72.9 to 82.3]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 84.0 [79.8 to 88.2] | 78.6 [73.9 to 83.2]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 82.7 [78.3 to 87.1] | 78.9 [74.1 to 83.6]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 79.4 [74.8 to 84.0] | 84.7 [80.5 to 88.9]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 80.7 [76.1 to 85.2] | 82.6 [78.2 to 87.0]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 78.9 [74.2 to 83.6] | 81.5 [77.0 to 86.0]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 81.3 [76.8 to 85.8] | 81.1 [76.5 to 85.7]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 80.5 [76.0 to 85.1] | 80.4 [75.8 to 85.0]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 79.5 [74.8 to 84.1] | 78.8 [74.0 to 83.6]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 81.0 [76.4 to 85.6] | 79.8 [75.2 to 84.5]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 80.0 [75.3 to 84.7] | 76.0 [71.0 to 81.1]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 78.7 [73.9 to 83.5] | 81.0 [76.3 to 85.7]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 78.7 [73.9 to 83.5] | 80.6 [75.9 to 85.4]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 81.3 [76.7 to 85.8] | 76.3 [71.2 to 81.4]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 76.3 [71.3 to 81.3] | 77.5 [72.5 to 82.6]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 75.7 [70.8 to 80.7] | 74.8 [69.6 to 80.0]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 76.6 [71.6 to 81.6] | 79.0 [74.0 to 84.0]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 78.8 [74.0 to 83.6] | 76.9 [71.7 to 82.1]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 74.6 [69.5 to 79.8] | 77.4 [72.3 to 82.5]

10. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 302 | 291
Percentage of participants
  Avoiding a Loss of ≥15 Letters | 95.8 [93.6 to 98.0] | 97.3 [95.5 to 99.1]
  Avoiding a Loss of ≥10 Letters | 93.8 [91.1 to 96.4] | 94.6 [92.2 to 97.1]
  Avoiding a Loss of ≥5 Letters | 91.2 [88.0 to 94.3] | 88.5 [85.0 to 92.0]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Avoiding a Loss of ≥15 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -1.5, 95% CI 2-sided [-4.4 to 1.3] — The treatment difference in CMH weighted percentage of participants avoiding a loss of ≥15 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 2: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Avoiding a Loss of ≥10 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -0.9, 95% CI 2-sided [-4.5 to 2.8] — The treatment difference in CMH weighted percentage of participants avoiding a loss of ≥10 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 3: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Avoiding a Loss of ≥5 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 2.6, 95% CI 2-sided [-2.1 to 7.3] — The treatment difference in CMH weighted percentage of participants avoiding a loss of ≥5 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

11. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 10
Time Frame: Baseline, average of Weeks 52, 56, and 60
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 289 | 276
Percentage of participants | 96.5 [94.4 to 98.6] | 96.1 [94.0 to 98.3]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 52-60; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-2.6 to 3.3] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters From the Baseline BCVA in the Study Eye Over Time
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The weighted percentage of participants avoiding a loss of letters in BCVA from baseline was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 99.4 [98.6 to 100.0] | 98.1 [96.7 to 99.6]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 98.5 [97.3 to 99.8] | 97.8 [96.3 to 99.4]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 98.5 [97.3 to 99.8] | 98.1 [96.7 to 99.6]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 97.6 [96.0 to 99.2] | 98.4 [97.0 to 99.8]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 97.3 [95.5 to 99.0] | 98.4 [97.0 to 99.7]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 96.6 [94.6 to 98.6] | 97.2 [95.4 to 99.1]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 97.0 [95.1 to 98.9] | 97.8 [96.2 to 99.5]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 97.0 [95.1 to 98.9] | 96.9 [95.0 to 98.9]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 97.0 [95.2 to 98.9] | 96.5 [94.5 to 98.6]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 96.2 [94.1 to 98.4] | 97.6 [95.9 to 99.3]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 95.9 [93.6 to 98.1] | 96.4 [94.3 to 98.5]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 95.8 [93.5 to 98.0] | 96.9 [95.0 to 98.8]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 94.9 [92.5 to 97.4] | 96.8 [94.8 to 98.8]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 96.1 [93.9 to 98.3] | 96.8 [94.8 to 98.8]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 95.0 [92.5 to 97.5] | 96.1 [94.0 to 98.3]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 96.4 [94.3 to 98.5] | 94.9 [92.3 to 97.4]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 94.7 [92.1 to 97.2] | 96.0 [93.7 to 98.3]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 94.5 [91.9 to 97.2] | 95.4 [92.9 to 97.9]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 94.9 [92.3 to 97.4] | 93.7 [90.9 to 96.6]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 93.9 [91.1 to 96.6] | 93.3 [90.4 to 96.3]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 92.5 [89.5 to 95.5] | 93.8 [90.9 to 96.7]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 94.1 [91.4 to 96.7] | 94.3 [91.5 to 97.0]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 93.0 [90.2 to 95.9] | 94.6 [92.0 to 97.2]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 92.6 [89.6 to 95.6] | 95.0 [92.5 to 97.6]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 92.5 [89.5 to 95.5] | 93.9 [91.1 to 96.7]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 92.9 [90.0 to 95.9] | 94.0 [91.0 to 96.9]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 92.3 [89.2 to 95.3] | 93.3 [90.3 to 96.3]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 91.8 [88.7 to 95.0] | 93.0 [89.9 to 96.1]

13. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥10 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 12
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 98.5 [97.2 to 99.8] | 96.2 [94.1 to 98.3]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 97.0 [95.3 to 98.7] | 96.9 [95.0 to 98.7]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 97.0 [95.2 to 98.8] | 96.8 [94.9 to 98.7]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 96.6 [94.7 to 98.5] | 96.8 [94.9 to 98.7]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 95.2 [92.9 to 97.4] | 96.1 [94.0 to 98.2]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 95.2 [92.9 to 97.6] | 95.5 [93.2 to 97.8]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 95.0 [92.6 to 97.4] | 95.2 [92.7 to 97.7]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 94.6 [92.1 to 97.1] | 95.9 [93.7 to 98.1]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 95.3 [93.0 to 97.7] | 94.4 [91.8 to 97.0]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 93.8 [91.1 to 96.5] | 94.6 [92.2 to 97.1]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 94.1 [91.4 to 96.8] | 92.1 [89.1 to 95.1]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 92.2 [89.2 to 95.3] | 94.8 [92.3 to 97.3]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 91.4 [88.2 to 94.6] | 93.8 [91.1 to 96.6]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 93.3 [90.5 to 96.2] | 95.0 [92.5 to 97.5]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 91.4 [88.2 to 94.6] | 93.2 [90.4 to 96.1]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 93.5 [90.7 to 96.4] | 92.3 [89.3 to 95.4]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 91.9 [88.8 to 95.0] | 92.9 [89.9 to 96.0]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 92.4 [89.3 to 95.5] | 91.6 [88.3 to 94.9]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 93.1 [90.2 to 96.0] | 90.1 [86.5 to 93.6]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 92.1 [89.0 to 95.2] | 89.9 [86.3 to 93.5]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 90.3 [86.9 to 93.7] | 91.8 [88.4 to 95.1]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 90.8 [87.5 to 94.1] | 92.3 [89.1 to 95.4]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 90.7 [87.4 to 94.1] | 91.0 [87.6 to 94.5]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 90.4 [87.0 to 93.8] | 92.6 [89.4 to 95.8]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 90.7 [87.4 to 94.0] | 91.6 [88.3 to 94.9]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 89.0 [85.4 to 92.7] | 92.2 [88.9 to 95.4]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 88.5 [84.8 to 92.3] | 91.2 [87.7 to 94.7]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 88.5 [84.7 to 92.2] | 89.5 [85.8 to 93.2]

14. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥5 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 12
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 93.0 [90.4 to 95.6] | 91.8 [88.9 to 94.7]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 93.1 [90.4 to 95.7] | 94.1 [91.5 to 96.6]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 93.3 [90.7 to 95.9] | 91.8 [88.8 to 94.7]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 91.7 [88.7 to 94.6] | 90.8 [87.7 to 94.0]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 92.0 [89.1 to 94.9] | 92.9 [90.0 to 95.7]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 90.6 [87.4 to 93.9] | 91.7 [88.6 to 94.8]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 91.0 [87.9 to 94.1] | 90.2 [86.7 to 93.7]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 89.9 [86.5 to 93.2] | 91.0 [87.7 to 94.3]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 90.7 [87.5 to 94.0] | 87.4 [83.6 to 91.2]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 91.7 [88.6 to 94.9] | 88.1 [84.5 to 91.7]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 90.9 [87.7 to 94.2] | 88.8 [85.3 to 92.3]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 89.4 [85.9 to 93.0] | 88.6 [85.0 to 92.2]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 88.9 [85.3 to 92.5] | 91.7 [88.6 to 94.8]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 89.5 [86.0 to 93.0] | 88.8 [85.2 to 92.5]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 86.7 [82.9 to 90.6] | 88.8 [85.2 to 92.4]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 87.8 [84.1 to 91.6] | 86.0 [82.0 to 90.1]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 88.2 [84.5 to 91.9] | 87.1 [83.2 to 91.0]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 87.0 [83.1 to 90.9] | 87.3 [83.4 to 91.2]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 87.1 [83.2 to 91.1] | 85.4 [81.2 to 89.5]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 87.3 [83.5 to 91.2] | 82.8 [78.3 to 87.3]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 84.1 [79.9 to 88.4] | 87.1 [83.1 to 91.2]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 87.5 [83.7 to 91.3] | 86.6 [82.5 to 90.6]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 87.0 [83.1 to 90.9] | 87.2 [83.2 to 91.2]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 82.7 [78.4 to 87.1] | 86.2 [82.1 to 90.4]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 85.9 [81.9 to 89.8] | 84.2 [79.9 to 88.5]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 83.5 [79.1 to 87.8] | 85.4 [81.1 to 89.7]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 84.1 [79.9 to 88.4] | 83.9 [79.4 to 88.5]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 82.2 [77.7 to 86.7] | 84.4 [80.0 to 88.8]

15. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: as for outcome 4
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 302 | 291
Percentage of participants | 24.5 [19.8 to 29.2] | 26.2 [21.2 to 31.1]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -1.7, 95% CI 2-sided [-8.5 to 5.1] — The treatment difference in CMH weighted percentage of participants gaining ≥15 letters or achieving BCVA ≥84 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

16. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 11.3 [7.9 to 14.6] | 12.4 [8.9 to 15.9]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 16.5 [12.5 to 20.4] | 16.1 [12.2 to 20.0]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 22.0 [17.7 to 26.4] | 21.1 [16.7 to 25.4]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 21.7 [17.4 to 26.1] | 20.7 [16.2 to 25.1]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 24.9 [20.2 to 29.5] | 24.9 [20.2 to 29.6]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 23.6 [18.9 to 28.3] | 23.7 [18.9 to 28.6]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 27.7 [22.7 to 32.7] | 26.9 [21.8 to 32.1]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 28.7 [23.6 to 33.8] | 23.2 [18.4 to 27.9]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 25.9 [21.1 to 30.7] | 24.6 [19.7 to 29.5]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 27.9 [22.9 to 32.9] | 31.1 [25.9 to 36.4]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 27.2 [22.2 to 32.1] | 28.1 [22.8 to 33.3]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 27.3 [22.3 to 32.4] | 28.3 [23.1 to 33.6]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 29.2 [24.1 to 34.3] | 28.3 [23.1 to 33.5]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 32.0 [26.7 to 37.2] | 31.5 [26.1 to 36.9]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 27.5 [22.5 to 32.5] | 31.4 [26.0 to 36.8]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 30.1 [25.0 to 35.3] | 27.1 [21.9 to 32.3]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 28.3 [23.1 to 33.4] | 30.0 [24.6 to 35.3]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 26.4 [21.4 to 31.4] | 31.5 [26.0 to 36.9]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 27.4 [22.2 to 32.5] | 29.2 [23.9 to 34.4]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 28.7 [23.4 to 34.0] | 31.2 [25.7 to 36.6]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 28.0 [22.8 to 33.1] | 30.1 [24.6 to 35.5]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 29.1 [23.8 to 34.4] | 28.4 [23.2 to 33.6]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 27.0 [21.8 to 32.1] | 29.0 [23.6 to 34.3]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 30.7 [25.3 to 36.0] | 31.1 [25.5 to 36.6]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 28.6 [23.3 to 33.9] | 27.2 [22.0 to 32.5]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 27.2 [22.0 to 32.4] | 30.2 [24.8 to 35.6]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 26.3 [21.1 to 31.4] | 27.0 [21.7 to 32.4]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 29.4 [24.1 to 34.7] | 26.5 [21.4 to 31.6]

17. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (<69 letters vs. ≥69 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 302 | 291
Percentage of participants | 55.2 [50.1 to 60.2] | 49.4 [44.4 to 54.4]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 5.7, 95% CI 2-sided [-1.4 to 12.9] — The treatment difference in CMH weighted percentage of participants achieving BCVA ≥69 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

18. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Over Time
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (<69 letters vs. ≥69 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 45.7 [41.1 to 50.2] | 40.1 [35.8 to 44.5]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 50.5 [45.8 to 55.1] | 45.2 [40.7 to 49.7]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 53.5 [48.8 to 58.3] | 48.5 [43.8 to 53.3]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 56.1 [51.2 to 60.9] | 47.4 [42.8 to 52.1]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 57.5 [52.6 to 62.4] | 51.1 [46.3 to 55.9]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 57.4 [52.4 to 62.4] | 47.8 [42.9 to 52.8]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 55.2 [50.0 to 60.4] | 48.2 [43.2 to 53.2]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 55.9 [50.8 to 61.1] | 49.8 [45.0 to 54.6]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 56.0 [50.9 to 61.0] | 47.4 [42.2 to 52.6]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 54.7 [49.5 to 59.9] | 52.7 [47.5 to 57.9]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 56.3 [51.4 to 61.3] | 52.5 [47.3 to 57.7]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 55.0 [49.8 to 60.2] | 52.3 [47.1 to 57.5]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 55.9 [50.6 to 61.1] | 55.6 [50.4 to 60.9]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 57.1 [51.8 to 62.3] | 52.9 [47.7 to 58.2]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 53.0 [47.6 to 58.3] | 53.6 [48.3 to 58.9]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 58.8 [53.5 to 64.2] | 52.9 [47.5 to 58.3]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 57.0 [51.7 to 62.4] | 55.5 [50.0 to 60.9]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 58.1 [52.7 to 63.4] | 53.3 [48.0 to 58.6]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 58.0 [52.6 to 63.4] | 54.0 [48.6 to 59.3]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 57.3 [52.0 to 62.6] | 51.9 [46.5 to 57.4]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 58.4 [53.1 to 63.7] | 56.9 [51.5 to 62.4]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 57.2 [51.9 to 62.6] | 51.1 [45.6 to 56.5]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 56.1 [50.8 to 61.4] | 54.9 [49.5 to 60.3]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 55.5 [49.9 to 61.0] | 53.9 [48.4 to 59.4]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 55.1 [49.5 to 60.7] | 51.7 [46.2 to 57.2]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 55.1 [49.4 to 60.7] | 52.8 [47.3 to 58.2]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 54.8 [49.1 to 60.4] | 51.0 [45.5 to 56.5]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 55.7 [50.2 to 61.1] | 51.0 [45.6 to 56.4]

19. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: as for outcome 4
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 302 | 291
Percentage of participants | 7.9 [5.0 to 10.8] | 7.5 [4.7 to 10.3]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 0.4, 95% CI 2-sided [-3.6 to 4.4] — The treatment difference in CMH weighted percentage of participants with BCVA ≤38 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

20. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 328 | 323
  Week 4 | 6.8 [4.3 to 9.4] | 6.1 [3.7 to 8.5]
  Week 8: number analyzed (Participants) | 327 | 322
  Week 8 | 7.4 [4.8 to 10.1] | 6.2 [3.7 to 8.6]
  Week 12: number analyzed (Participants) | 326 | 317
  Week 12 | 7.6 [5.0 to 10.2] | 5.9 [3.5 to 8.3]
  Week 16: number analyzed (Participants) | 321 | 315
  Week 16 | 9.5 [6.6 to 12.5] | 5.3 [3.0 to 7.6]
  Week 20: number analyzed (Participants) | 320 | 309
  Week 20 | 9.3 [6.4 to 12.3] | 5.7 [3.3 to 8.1]
  Week 24: number analyzed (Participants) | 295 | 288
  Week 24 | 8.1 [5.2 to 11.1] | 6.3 [3.7 to 8.9]
  Week 28: number analyzed (Participants) | 292 | 271
  Week 28 | 7.4 [4.6 to 10.3] | 6.4 [3.7 to 9.1]
  Week 32: number analyzed (Participants) | 287 | 288
  Week 32 | 8.1 [5.1 to 11.0] | 6.6 [4.0 to 9.2]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 7.8 [4.9 to 10.6] | 6.8 [4.1 to 9.5]
  Week 40: number analyzed (Participants) | 286 | 288
  Week 40 | 8.3 [5.3 to 11.3] | 7.6 [4.8 to 10.3]
  Week 44: number analyzed (Participants) | 285 | 273
  Week 44 | 7.9 [4.9 to 10.9] | 6.8 [4.0 to 9.5]
  Week 48: number analyzed (Participants) | 282 | 277
  Week 48 | 9.7 [6.5 to 12.9] | 6.3 [3.6 to 9.0]
  Week 52: number analyzed (Participants) | 283 | 273
  Week 52 | 9.1 [6.0 to 12.2] | 6.5 [3.7 to 9.2]
  Week 56: number analyzed (Participants) | 283 | 273
  Week 56 | 8.1 [5.1 to 11.1] | 6.3 [3.6 to 9.0]
  Week 60: number analyzed (Participants) | 278 | 273
  Week 60 | 8.2 [5.2 to 11.3] | 7.3 [4.5 to 10.2]
  Week 64: number analyzed (Participants) | 276 | 266
  Week 64 | 7.1 [4.2 to 10.1] | 7.2 [4.3 to 10.1]
  Week 68: number analyzed (Participants) | 276 | 266
  Week 68 | 8.8 [5.6 to 12.0] | 6.8 [4.0 to 9.6]
  Week 72: number analyzed (Participants) | 276 | 261
  Week 72 | 8.4 [5.2 to 11.6] | 6.2 [3.4 to 8.9]
  Week 76: number analyzed (Participants) | 268 | 267
  Week 76 | 9.5 [6.2 to 12.9] | 7.4 [4.5 to 10.3]
  Week 80: number analyzed (Participants) | 275 | 264
  Week 80 | 9.8 [6.5 to 13.1] | 8.4 [5.3 to 11.5]
  Week 84: number analyzed (Participants) | 279 | 254
  Week 84 | 9.3 [6.0 to 12.6] | 7.2 [4.2 to 10.1]
  Week 88: number analyzed (Participants) | 276 | 253
  Week 88 | 8.4 [5.2 to 11.6] | 7.5 [4.5 to 10.4]
  Week 92: number analyzed (Participants) | 273 | 253
  Week 92 | 8.9 [5.6 to 12.2] | 9.0 [5.8 to 12.2]
  Week 96: number analyzed (Participants) | 266 | 247
  Week 96 | 10.4 [6.8 to 13.9] | 9.7 [6.5 to 13.0]
  Week 100: number analyzed (Participants) | 272 | 254
  Week 100 | 10.3 [6.8 to 13.8] | 10.9 [7.5 to 14.4]
  Week 104: number analyzed (Participants) | 263 | 249
  Week 104 | 9.2 [5.8 to 12.6] | 9.8 [6.4 to 13.1]
  Week 108: number analyzed (Participants) | 267 | 247
  Week 108 | 9.5 [6.0 to 12.9] | 10.0 [6.5 to 13.4]
  Week 112: number analyzed (Participants) | 267 | 254
  Week 112 | 9.0 [5.7 to 12.4] | 10.6 [7.1 to 14.0]

21. Secondary Outcome: Percentage of Participants in the Faricimab Arm on Once Every 8-Weeks, 12-Weeks, or 16-Weeks Treatment Intervals Among Those Completing Week 48
Description: Percentages are based on the number of participants randomized to the faricimab arm who have not discontinued the study at Week 48. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit. The 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Week 48
Population: The analysis included all participants randomized to the faricimab arm who completed their Week 48 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 316
Percentage of participants
  Once Every 8 Weeks | 22.2 [17.6 to 26.7]
  Once Every 12 Weeks | 32.9 [27.7 to 38.1]
  Once Every 16 Weeks | 44.9 [39.4 to 50.4]

22. Secondary Outcome: Percentage of Participants in the Faricimab Arm on Once Every 8-Weeks, 12-Weeks, or 16-Weeks Treatment Intervals Among Those Completing Week 60
Description: Percentages are based on the number of participants randomized to the faricimab arm who have not discontinued the study at Week 60. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit. The 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Week 60
Population: The analysis included all participants randomized to the faricimab arm who completed their Week 60 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 305
Percentage of participants
  Once Every 8 Weeks | 21.6 [17.0 to 26.3]
  Once Every 12 Weeks | 32.8 [27.5 to 38.1]
  Once Every 16 Weeks | 45.6 [40.0 to 51.2]

23. Secondary Outcome: Percentage of Participants in the Faricimab Arm on Once Every 8-Weeks, 12-Weeks, or 16-Weeks Treatment Intervals Among Those Completing Week 112
Description: Percentages are based on the number of participants randomized to the faricimab arm who have not discontinued the study at Week 112. Treatment interval at a given visit is defined as the treatment interval decision followed at that visit. Treatment interval at Week 112 is calculated using data recorded at Week 108. The 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Weeks 108 and 112
Population: The analysis included all participants randomized to the faricimab arm who completed their Week 112 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 287
Percentage of participants
  Once Every 8 Weeks | 18.8 [14.3 to 23.3]
  Once Every 12 Weeks | 14.3 [10.2 to 18.3]
  Once Every 16 Weeks | 66.9 [61.4 to 72.4]

24. Secondary Outcome: Number of Study Drug Injections Received in the Study Eye Through Week 48
Time Frame: From Baseline through Week 48
Population: Safety Evaluable Population: all participants who received at least one dose of active study drug (faricimab or aflibercept) in the study eye.
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 326
Injections | 6.0 [1 to 8] | 8.0 [1 to 8]

25. Secondary Outcome: Number of Study Drug Injections Received in the Study Eye Through Week 60
Time Frame: From Baseline through Week 60
Population: as for outcome 24
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 326
Injections | 7.0 [1 to 10] | 9.0 [1 to 9]

26. Secondary Outcome: Number of Study Drug Injections Received in the Study Eye Through Week 108
Time Frame: From Baseline through Week 108
Population: as for outcome 24
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 326
Injections | 10.0 [1 to 16] | 15.0 [1 to 15]

27. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using optical coherence tomography (OCT), as assessed by the central reading center. For the Mixed Model of Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group iteraction, baseline CST (continuous), baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (<33 letters and ≥33 letters), and region (U.S. and Canada, Asia, and the rest of the world). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
microns | -137.1 [-143.1 to -131.2] | -130.8 [-136.8 to -124.8]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in Adjusted Means at Weeks 40-48; Test type: Other; Adjusted mean difference = -6.4, 95% CI 2-sided [-14.8 to 2.1], Standard Error of Mean 4.30 — The treatment difference in adjusted means of change from baseline CST is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept. MMRM adjustments are listed in the outcome measure description

28. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using optical coherence tomography (OCT), as assessed by the central reading center. For the Mixed Model of Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline CST (continuous), baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (<33 letters and ≥33 letters), and region (U.S. and Canada, Asia, and the rest of the world). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 60
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
microns | -135.7 [-141.2 to -130.1] | -137.0 [-142.7 to -131.3]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in Adjusted Means at Weeks 52-60; Test type: Other; Adjusted mean difference = 1.4, 95% CI 2-sided [-6.6 to 9.3], Standard Error of Mean 4.05 — [estimate comment as in outcome 27, analysis 1]

29. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Over Time
Description: as for outcome 28
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
microns
  Week 4 | -126.5 [-132.3 to -120.6] | -113.9 [-119.8 to -108.0]
  Week 8 | -138.0 [-143.7 to -132.3] | -123.8 [-129.6 to -118.0]
  Week 12 | -141.7 [-147.1 to -136.3] | -129.6 [-135.0 to -124.1]
  Week 16 | -143.7 [-150.3 to -137.1] | -112.9 [-119.6 to -106.2]
  Week 20 | -130.9 [-136.8 to -125.0] | -132.9 [-138.8 to -126.9]
  Week 24 | -130.1 [-137.1 to -123.1] | -112.2 [-119.3 to -105.2]
  Week 28 | -127.3 [-134.0 to -120.6] | -130.1 [-136.9 to -123.3]
  Week 32 | -138.6 [-145.8 to -131.5] | -115.3 [-122.5 to -108.1]
  Week 36 | -124.6 [-131.3 to -118.0] | -135.2 [-141.9 to -128.5]
  Week 40 | -142.5 [-149.3 to -135.6] | -122.5 [-129.4 to -115.6]
  Week 44 | -130.9 [-136.7 to -125.1] | -141.6 [-147.6 to -135.7]
  Week 48 | -135.5 [-142.3 to -128.6] | -123.9 [-130.8 to -117.0]
  Week 52 | -140.9 [-146.4 to -135.3] | -139.6 [-145.3 to -134.0]
  Week 56 | -138.9 [-145.7 to -132.1] | -125.6 [-132.5 to -118.6]
  Week 60 | -125.9 [-132.0 to -119.7] | -142.3 [-148.6 to -136.1]
  Week 64 | -143.8 [-150.3 to -137.2] | -126.0 [-132.7 to -119.3]
  Week 68 | -138.0 [-143.9 to -132.2] | -138.8 [-144.8 to -132.8]
  Week 72 | -140.7 [-147.3 to -134.1] | -128.8 [-135.5 to -122.0]
  Week 76 | -136.1 [-142.4 to -129.7] | -139.0 [-145.4 to -132.6]
  Week 80 | -144.4 [-151.1 to -137.8] | -128.7 [-135.5 to -121.9]
  Week 84 | -143.5 [-149.2 to -137.8] | -143.2 [-149.1 to -137.4]
  Week 88 | -145.5 [-151.6 to -139.5] | -133.3 [-139.5 to -127.1]
  Week 92 | -142.1 [-148.0 to -136.1] | -143.2 [-149.3 to -137.1]
  Week 96 | -146.8 [-153.1 to -140.4] | -134.7 [-141.2 to -128.2]
  Week 100 | -145.0 [-151.7 to -138.3] | -146.2 [-153.1 to -139.3]
  Week 104 | -149.6 [-156.3 to -142.8] | -137.4 [-144.3 to -130.5]
  Week 108 | -148.5 [-154.4 to -142.6] | -148.3 [-154.4 to -142.2]
  Week 112 | -152.9 [-159.2 to -146.7] | -139.1 [-145.5 to -132.7]

30. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye Over Time
Description: Intraretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 millimetre [mm]). The weighted estimates of the percentage of participants with absence of intraretinal fluid were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 324 | 320
  Week 4 | 86.9 [83.5 to 90.4] | 82.9 [78.9 to 87.0]
  Week 8: number analyzed (Participants) | 324 | 316
  Week 8 | 88.5 [85.2 to 91.9] | 84.6 [80.7 to 88.5]
  Week 12: number analyzed (Participants) | 323 | 315
  Week 12 | 87.5 [84.0 to 91.0] | 84.5 [80.6 to 88.5]
  Week 16: number analyzed (Participants) | 320 | 314
  Week 16 | 90.6 [87.5 to 93.7] | 76.5 [71.9 to 81.0]
  Week 20: number analyzed (Participants) | 320 | 305
  Week 20 | 78.8 [74.5 to 83.0] | 86.1 [82.3 to 89.8]
  Week 24: number analyzed (Participants) | 294 | 284
  Week 24 | 78.7 [74.2 to 83.1] | 78.0 [73.4 to 82.7]
  Week 28: number analyzed (Participants) | 291 | 273
  Week 28 | 77.1 [72.4 to 81.8] | 85.9 [81.8 to 89.9]
  Week 32: number analyzed (Participants) | 286 | 291
  Week 32 | 86.3 [82.5 to 90.2] | 78.3 [73.6 to 82.9]
  Week 36: number analyzed (Participants) | 293 | 278
  Week 36 | 79.6 [75.0 to 84.1] | 86.1 [82.1 to 90.1]
  Week 40: number analyzed (Participants) | 277 | 278
  Week 40 | 84.5 [80.3 to 88.7] | 77.5 [72.7 to 82.3]
  Week 44: number analyzed (Participants) | 275 | 258
  Week 44 | 78.5 [73.7 to 83.2] | 84.2 [79.9 to 88.5]
  Week 48: number analyzed (Participants) | 274 | 269
  Week 48 | 84.1 [79.8 to 88.4] | 77.7 [72.8 to 82.5]
  Week 52: number analyzed (Participants) | 281 | 270
  Week 52 | 85.9 [81.9 to 89.8] | 85.3 [81.1 to 89.4]
  Week 56: number analyzed (Participants) | 281 | 272
  Week 56 | 85.2 [81.1 to 89.2] | 81.1 [76.6 to 85.6]
  Week 60: number analyzed (Participants) | 273 | 266
  Week 60 | 77.8 [73.0 to 82.6] | 85.4 [81.2 to 89.5]
  Week 104: number analyzed (Participants) | 259 | 247
  Week 104 | 86.0 [81.9 to 90.1] | 80.0 [75.1 to 84.9]
  Week 108: number analyzed (Participants) | 264 | 243
  Week 108 | 82.2 [77.7 to 86.6] | 83.5 [79.0 to 88.1]
  Week 112: number analyzed (Participants) | 266 | 251
  Week 112 | 85.9 [81.8 to 90.0] | 80.5 [75.7 to 85.4]

31. Secondary Outcome: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye Over Time
Description: Subretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants with absence of subretinal fluid were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 319
  Week 4 | 70.9 [66.1 to 75.7] | 61.7 [56.4 to 66.9]
  Week 8: number analyzed (Participants) | 323 | 319
  Week 8 | 79.8 [75.6 to 84.1] | 73.6 [68.9 to 78.4]
  Week 12: number analyzed (Participants) | 324 | 315
  Week 12 | 88.6 [85.1 to 92.0] | 79.6 [75.3 to 84.0]
  Week 16: number analyzed (Participants) | 320 | 315
  Week 16 | 90.6 [87.4 to 93.8] | 63.8 [58.6 to 68.9]
  Week 20: number analyzed (Participants) | 320 | 308
  Week 20 | 76.1 [71.6 to 80.7] | 80.4 [76.1 to 84.8]
  Week 24: number analyzed (Participants) | 295 | 287
  Week 24 | 73.7 [68.8 to 78.5] | 59.1 [53.5 to 64.6]
  Week 28: number analyzed (Participants) | 292 | 272
  Week 28 | 71.5 [66.6 to 76.4] | 78.7 [73.9 to 83.5]
  Week 32: number analyzed (Participants) | 287 | 291
  Week 32 | 82.6 [78.3 to 87.0] | 62.2 [56.7 to 67.7]
  Week 36: number analyzed (Participants) | 293 | 282
  Week 36 | 70.6 [65.5 to 75.7] | 80.7 [76.1 to 85.2]
  Week 40: number analyzed (Participants) | 283 | 285
  Week 40 | 77.6 [72.9 to 82.3] | 63.9 [58.4 to 69.5]
  Week 44: number analyzed (Participants) | 280 | 269
  Week 44 | 65.7 [60.3 to 71.0] | 76.2 [71.1 to 81.2]
  Week 48: number analyzed (Participants) | 278 | 274
  Week 48 | 72.5 [67.5 to 77.5] | 62.1 [56.5 to 67.7]
  Week 52: number analyzed (Participants) | 281 | 271
  Week 52 | 83.0 [78.8 to 87.3] | 80.6 [76.0 to 85.3]
  Week 56: number analyzed (Participants) | 282 | 271
  Week 56 | 80.7 [76.3 to 85.2] | 71.6 [66.4 to 76.8]
  Week 60: number analyzed (Participants) | 278 | 271
  Week 60 | 63.6 [58.1 to 69.0] | 80.0 [75.3 to 84.8]
  Week 104: number analyzed (Participants) | 262 | 248
  Week 104 | 80.0 [75.3 to 84.7] | 73.9 [68.5 to 79.3]
  Week 108: number analyzed (Participants) | 266 | 244
  Week 108 | 76.1 [71.2 to 81.0] | 80.7 [75.8 to 85.5]
  Week 112: number analyzed (Participants) | 267 | 252
  Week 112 | 80.9 [76.4 to 85.4] | 77.5 [72.4 to 82.6]

32. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye Over Time
Description: Intraretinal fluid and subretinal fluid were measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants with absence of intraretinal and subretinal fluid were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 324 | 319
  Week 4 | 59.5 [54.2 to 64.8] | 49.8 [44.4 to 55.2]
  Week 8: number analyzed (Participants) | 323 | 315
  Week 8 | 70.2 [65.2 to 75.1] | 61.6 [56.3 to 66.9]
  Week 12: number analyzed (Participants) | 323 | 315
  Week 12 | 77.0 [72.4 to 81.5] | 66.6 [61.5 to 71.7]
  Week 16: number analyzed (Participants) | 319 | 315
  Week 16 | 82.4 [78.3 to 86.5] | 47.6 [42.2 to 53.0]
  Week 20: number analyzed (Participants) | 320 | 305
  Week 20 | 62.3 [57.3 to 67.4] | 68.6 [63.6 to 73.7]
  Week 24: number analyzed (Participants) | 295 | 284
  Week 24 | 56.5 [50.8 to 62.1] | 45.4 [39.7 to 51.1]
  Week 28: number analyzed (Participants) | 291 | 273
  Week 28 | 55.5 [49.9 to 61.1] | 66.5 [61.0 to 72.0]
  Week 32: number analyzed (Participants) | 286 | 291
  Week 32 | 73.1 [68.0 to 78.1] | 48.6 [42.9 to 54.3]
  Week 36: number analyzed (Participants) | 293 | 278
  Week 36 | 56.3 [50.8 to 61.9] | 68.3 [62.9 to 73.7]
  Week 40: number analyzed (Participants) | 278 | 281
  Week 40 | 65.8 [60.3 to 71.2] | 49.0 [43.2 to 54.8]
  Week 44: number analyzed (Participants) | 277 | 262
  Week 44 | 49.5 [43.7 to 55.3] | 64.3 [58.5 to 70.0]
  Week 48: number analyzed (Participants) | 277 | 270
  Week 48 | 62.2 [56.6 to 67.8] | 46.1 [40.3 to 52.0]
  Week 52: number analyzed (Participants) | 281 | 270
  Week 52 | 70.3 [65.2 to 75.5] | 68.8 [63.4 to 74.3]
  Week 56: number analyzed (Participants) | 281 | 272
  Week 56 | 66.9 [61.5 to 72.3] | 57.5 [51.8 to 63.3]
  Week 60: number analyzed (Participants) | 275 | 266
  Week 60 | 49.3 [43.5 to 55.0] | 69.1 [63.6 to 74.6]
  Week 104: number analyzed (Participants) | 259 | 247
  Week 104 | 68.1 [62.5 to 73.7] | 58.6 [52.7 to 64.6]
  Week 108: number analyzed (Participants) | 264 | 243
  Week 108 | 61.6 [55.9 to 67.3] | 67.1 [61.3 to 72.9]
  Week 112: number analyzed (Participants) | 266 | 251
  Week 112 | 68.7 [63.3 to 74.1] | 61.1 [55.1 to 67.1]

33. Secondary Outcome: Percentage of Participants With Absence of Pigment Epithelial Detachment in the Study Eye Over Time
Description: Pigment epithelial detachment was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants with absence of pigment epithelial detachment were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 327
Percentage of participants
  Week 4: number analyzed (Participants) | 323 | 320
  Week 4 | 3.7 [1.7 to 5.8] | 5.6 [3.1 to 8.1]
  Week 8: number analyzed (Participants) | 321 | 318
  Week 8 | 3.1 [1.3 to 5.0] | 4.1 [1.9 to 6.2]
  Week 12: number analyzed (Participants) | 321 | 314
  Week 12 | 4.7 [2.4 to 7.0] | 5.5 [3.0 to 8.0]
  Week 16: number analyzed (Participants) | 316 | 313
  Week 16 | 2.5 [0.8 to 4.1] | 5.8 [3.2 to 8.4]
  Week 20: number analyzed (Participants) | 316 | 306
  Week 20 | 3.8 [1.7 to 5.9] | 6.0 [3.4 to 8.6]
  Week 24: number analyzed (Participants) | 293 | 284
  Week 24 | 4.1 [1.8 to 6.3] | 4.9 [2.5 to 7.4]
  Week 28: number analyzed (Participants) | 292 | 273
  Week 28 | 2.6 [0.9 to 4.4] | 1.9 [0.3 to 3.5]
  Week 32: number analyzed (Participants) | 287 | 291
  Week 32 | 4.3 [2.0 to 6.6] | 1.8 [0.3 to 3.3]
  Week 36: number analyzed (Participants) | 293 | 283
  Week 36 | 4.8 [2.4 to 7.1] | 3.9 [1.7 to 6.1]
  Week 40: number analyzed (Participants) | 284 | 286
  Week 40 | 6.3 [3.5 to 9.0] | 7.3 [4.4 to 10.3]
  Week 44: number analyzed (Participants) | 282 | 270
  Week 44 | 3.9 [1.7 to 6.2] | 9.1 [5.9 to 12.4]
  Week 48: number analyzed (Participants) | 280 | 275
  Week 48 | 3.3 [1.2 to 5.3] | 6.5 [3.7 to 9.3]
  Week 52: number analyzed (Participants) | 273 | 267
  Week 52 | 5.8 [3.1 to 8.5] | 8.1 [5.0 to 11.3]
  Week 56: number analyzed (Participants) | 272 | 266
  Week 56 | 4.7 [2.3 to 7.2] | 5.2 [2.7 to 7.7]
  Week 60: number analyzed (Participants) | 278 | 271
  Week 60 | 3.5 [1.4 to 5.6] | 6.3 [3.4 to 9.1]
  Week 104: number analyzed (Participants) | 260 | 246
  Week 104 | 8.0 [4.8 to 11.2] | 8.3 [5.0 to 11.7]
  Week 108: number analyzed (Participants) | 264 | 244
  Week 108 | 6.9 [3.9 to 10.0] | 8.0 [4.7 to 11.2]
  Week 112: number analyzed (Participants) | 264 | 248
  Week 112 | 8.1 [4.9 to 11.3] | 12.5 [8.4 to 16.5]

34. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Cysts in the Study Eye Over Time
Time Frame: Up to 112 weeks
Population: The percentage of participants with absence of intraretinal cysts over time was planned but it was not evaluated (i.e., 0 participants analyzed) because the absence of intraretinal fluid and the absence of intraretinal cysts are described by the same variable during reading center grading.
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Lesion in the Study Eye at Week 48
Description: The total area of the choroidal neovascularization lesion in the study eye was evaluated by a central reading center using fundus fluorescein angiography (FFA). Assessments were censored following COVID-19 related intercurrent events. Baseline was defined as the last available measurement obtained on or prior to randomization.
Time Frame: Baseline and Week 48
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and Week 48 were included in this analysis.
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 240 | 236
millimetres squared (mm^2) | 0.3 (4.6) | 1.1 (4.4)

36. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Lesion in the Study Eye at Week 112
Description: as for outcome 35
Time Frame: Baseline and Week 112
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and Week 112 were included in this analysis.
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 240 | 224
millimetres squared (mm^2) | 1.7 (7.5) | 1.7 (4.2)

37. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Leakage in the Study Eye at Week 48
Description: The total area of choroidal neovascularization leakage in the study eye was evaluated by a central reading center using fundus fluorescein angiography (FFA). Assessments were censored following COVID-19 related intercurrent events. Baseline was defined as the last available measurement obtained on or prior to randomization.
Time Frame: Baseline and Week 48
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 241 | 238
millimetres squared (mm^2) | -3.3 (6.6) | -2.1 (6.3)

38. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Leakage in the Study Eye at Week 112
Description: as for outcome 37
Time Frame: Baseline and Week 112
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 239 | 220
millimetres squared (mm^2) | -5.3 (7.2) | -4.2 (5.9)

39. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: This analysis of adverse events (AEs) includes both ocular and non-ocular (systemic) AEs. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. AEs of special interest included the following: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law; Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 326
Percentage of participants
  Adverse Event (AE) | 84.9 | 88.0
  Serious AE (SAE) | 27.5 | 31.0
  AE Leading to Withdrawal from Study Treatment | 4.8 | 2.8
  AE of Special Interest (AESI) | 7.3 | 6.1

40. Secondary Outcome: Percentage of Participants With at Least One Ocular Adverse Event in the Study Eye or the Fellow Eye
Description: This analysis of adverse events (AEs) only includes ocular AEs, which are categorized as having occurred either in the study eye or the fellow eye. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 326
Percentage of participants
  Study Eye: Adverse Event (AE) | 52.9 | 47.5
  Study Eye: Serious AE (SAE) | 4.5 | 4.9
  Study Eye: AE Leading to Withdrawal from Treatment | 3.3 | 1.8
  Study Eye: Treatment-related AE | 3.6 | 3.1
  Study Eye: Treatment-related SAE | 1.8 | 0.6
  Study Eye: AE of Special Interest (AESI) | 3.9 | 4.3
  Study Eye: AESI, Drop in VA Score ≥30 Letters | 2.7 | 3.1
  Study Eye: AESI, Associated with Severe IOI | 0.6 | 0.3
  Study Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 0.6 | 0.9
  Study Eye: Suspected Transmission of Infectious Agent by Study Drug | 0.0 | 0.3
  Fellow Eye: AE | 46.2 | 41.7
  Fellow Eye: SAE | 3.6 | 2.5
  Fellow Eye: AESI | 3.0 | 2.1
  Fellow Eye: AESI, Drop in VA Score ≥30 Letters | 2.1 | 1.8
  Fellow Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 0.9 | 0.3

41. Secondary Outcome: Percentage of Participants With at Least One Non-Ocular Adverse Event
Description: This analysis of adverse events (AEs) only includes non-ocular (systemic) AEs. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. The non-ocular AE of special interest was: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 331 | 326
Percentage of participants
  Adverse Event (AE) | 71.0 | 75.8
  Serious AE (SAE) | 21.8 | 26.4
  AE Leading to Withdrawal from Study Treatment | 1.5 | 0.9
  AE of Special Interest (AESI) | 0.3 | 0.0

42. Secondary Outcome: Plasma Concentration of Faricimab Over Time
Description: Faricimab concentration in plasma was determined using a validated immunoassay method.
Time Frame: Pre-dose at Baseline, Weeks 4, 16, 20, 48, 76, and 112
Population: This analysis only includes Arm A participants who received treatment with faricimab in the pharmacokinetic-evaluable population, which includes safety-evaluable participants with at least one plasma sample, provided sufficient dosing information (dose and dosing time) was available. The number of participants analyzed at a given timepoint includes those with an available plasma sample and dosing information at that timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 331
micrograms per millilitre (μg/mL)
  Baseline: number analyzed (Participants) | 321
  Baseline | 0.0000 (0.0001)
  Week 4: number analyzed (Participants) | 319
  Week 4 | 0.0287 (0.0209)
  Week 16: number analyzed (Participants) | 300
  Week 16 | 0.0333 (0.0250)
  Week 20: number analyzed (Participants) | 305
  Week 20 | 0.0046 (0.0051)
  Week 48: number analyzed (Participants) | 273
  Week 48 | 0.0149 (0.0185)
  Week 76: number analyzed (Participants) | 269
  Week 76 | 0.0053 (0.0117)
  Week 112: number analyzed (Participants) | 278
  Week 112 | 0.0119 (0.0149)

43. Secondary Outcome: Percentage of Participants Who Tested Positive for Treatment-Emergent Anti-Drug Antibodies Against Faricimab During the Study
Description: Anti-drug antibodies (ADAs) against fariciamb were detected in plasma using a validated bridging enzyme-linked immunosorbent assay (ELISA). The percentage of participants with treatment-emergent ADA-positive samples includes post-baseline evaluable participants with at least one treatment-induced (defined as having an ADA-negative sample or missing sample at baseline and any positive post-baseline sample) or treatment-boosted (defined as having an ADA-positive sample at baseline and any positive post-baseline sample with a titer that is equal to or greater than 4-fold baseline titer) ADA-positive sample during the study treatment period.
Time Frame: Pre-dose at Baseline, Weeks 4, 20, 48, 76, and 112
Population: The immunogenicity-analysis population includes all participants randomized to the faricimab arm with at least one determinant ADA assessment. Only those with at least one post-baseline ADA assessment were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 330
Percentage of participants
  Total Treatment-Emergent ADA-Positive | 16.1
  Treatment-Induced ADA-Positive | 16.1
  Treatment-Boosted ADA-Positive | 0.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For ocular AEs, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
All-Cause Mortality (participants affected / at risk) | 10/331 | 14/326
Serious Adverse Events (participants affected / at risk) | 91/331 | 101/326
Other Adverse Events (participants affected / at risk) | 178/331 | 165/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab (N=331) | Arm B: Aflibercept (N=326)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 6 (11)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 3 (4)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1)
Eye allergy (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 8 (8) | 4 (4)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal pigment epithelial tear (Eye disorders) | 2 (2) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 2 (2) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 3 (3) | 1 (1)
Vitritis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Chorioretinitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Endophthalmitis (Infections and infestations) | 2 (2) | 3 (3)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 6 (7)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 5 (5)
Viral uveitis (Infections and infestations) | 2 (2) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sarcomatoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcomatoid carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 5 (9)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Postictal paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (3)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Corneal opacity (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (2)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 1 (1)
Peripheral exudative haemorrhagic chorioretinopathy (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 7 (7)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab (N=331) | Arm B: Aflibercept (N=326)
Conjunctival haemorrhage (Eye disorders) | 35 (47) | 37 (72)
Neovascular age-related macular degeneration (Eye disorders) | 80 (103) | 62 (81)
Nasopharyngitis (Infections and infestations) | 27 (33) | 22 (25)
Cataract (Eye disorders) | 38 (55) | 26 (38)
Dry eye (Eye disorders) | 15 (27) | 21 (37)
Posterior capsule opacification (Eye disorders) | 15 (20) | 19 (23)
Vitreous detachment (Eye disorders) | 22 (29) | 21 (26)
Urinary tract infection (Infections and infestations) | 19 (23) | 29 (36)
Fall (Injury, poisoning and procedural complications) | 18 (20) | 22 (27)
Hypertension (Vascular disorders) | 15 (15) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03823300/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03823300/SAP_001.pdf